CLINICAL TRIAL: NCT03896776
Title: A Pragmatic Trial of Two Strategies for Implementing an Effective eHealth HIV Prevention Program (Keep It Up! 3.0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Boston Medical Center (Other); Weill Medical College of Cornell University (Other); Marquette University (Other)
Responsible Party: Principal Investigator, Brian Mustanski, Director, Institute for Sexual and Gender Minority Health and Wellbeing, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH118213 (NIH)
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: HIV/AIDS; Gonorrhea; Chlamydia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Based Organization (CBO) Delivery (Experimental): CBOs will be selected through a Request for Proposal (RFP) process. The RFP will describe research and KIU! delivery activities to be conducted as part of the study and allowable budget to carry out the activities. The RFP will ask CBOs to describe past experience providing HIV services for YMSM. Selected CBOs will recruit participants into the intervention and encourage participants to complete each session of intervention content at baseline, 6 Week Follow-up, and 12 Week Follow-up.
  Participants in the CBO delivery arm will receive baseline HIV and STI testing at a CBO. Participants will receive an at-home STI test kit at 12 Week Follow-up if testing is not provided at their CBO site.
  Interventions: Behavioral: Keep It Up! 3.0
- Direct to Consumer (DTC) Delivery (Experimental): In the DTC arm, participants will be recruited online via paid social media advertising (e.g., Facebook, Instagram). Advertisements will target placements by age, gender, sexual orientation, racial background, "likes" that are relevant to YMSM (e.g., local LGBT organizations, "out" celebrities), and location (i.e., target county). Dating/sex-seeking apps (e.g., Grindr) will also be used to recruit YMSM, using a similar advertising approach as social media. These online recruitment strategies will be supplemented by referrals from local organizations and participant registries, and snowball recruitment. Study staff at Northwestern University will manage this recruitment process and encourage participants to complete each session of intervention content at baseline, 6 Week Follow-up, and 12 Week Follow-up.
  Participants in the DTC delivery arm will receive at-home HIV and STI test kits at baseline. Participants will receive an at-home STI test kit at 12 Week Follow-up.
  Interventions: Behavioral: Keep It Up! 3.0

INTERVENTIONS:
Behavioral: Keep It Up! 3.0 — KIU! is an online HIV prevention intervention developed for high-risk young men who have sex with men (YMSM) who recently tested HIV negative. Content was developed in collaboration with YMSM-serving CBOs and subjected to usability testing with diverse YMSM. The Information-Motivation-Behavioral Skills model and eLearning principles guided development of highly interactive, engaging, and culturally relevant health messages. KIU! involves 7 modules completed across 3 sessions, totaling ~1 hour of main content, plus 2 booster sessions at 6- and 12-week follow-ups. Each module is based on a setting or situation relevant to YMSM (e.g., connecting to the gay community and meeting guys through apps), with developmentally appropriate behavior change content embedded. KIU! uses diverse delivery methods (e.g. videos, animation, games) to address HIV knowledge gaps, motivate safer behaviors, teach behavioral skills, and instill self-efficacy for preventive behaviors.
  Other Names: KIU! 3.0

SUMMARY:
This study evaluates and compares two implementation strategies of an online HIV prevention intervention: Strategy 1 in which community-based organizations apply, and are selected, for funding to deliver Keep It Up! through current HIV testing programs; and Strategy 2 which is a "direct-to-consumer" model where centralized staff at Northwestern University recruit participants nationally through online advertising campaigns and manage engagement.

DETAILED DESCRIPTION:
Substantial effort has gone into developing and testing the efficacy of eHealth HIV prevention interventions, but these interventions will not affect the spread of the epidemic unless implemented effectively to reach the most at-risk populations. Despite emerging evidence that eHealth approaches can be highly effective in reducing HIV risk or improving care engagement, implementation requirements do not fit within established strategies for public health scale up, leaving it an open question as to how to bring these programs into practice. To date, little to no implementation science has examined strategies to effectively scale up eHealth HIV prevention programs.

The overarching goal of this study is to address this need by developing and evaluating novel strategies for implementing eHealth HIV prevention programs. Keep It Up! (KIU!) is an online program proven to reduce HIV risk among diverse young men who have sex with men (YMSM). KIU! was designed for YMSM who just tested HIV negative to keep it up and maintain negative status by reducing risk and enacting protections. Strong evidence of effectiveness on behavioral (decreased condomless sex) and biomedical outcomes (reduced STI incidence) makes KIU! an ideal eHealth intervention for implementation research. Lessons learned from KIU! implementation will set the pathway for implementing the many HIV eHealth programs currently undergoing efficacy testing.

Implementation strategies need to be evaluated using rigorous research designs. Through formative research with community-based organizations (CBOs), health departments, the CDC, and researchers, the investigators have identified two pragmatic implementation strategies that will be evaluated and compared:

In Strategy 1, CBOs apply for, and are selected for, funding to deliver KIU! through current HIV testing programs. Because CBOs do not have the capacity to host the technology, KIU! is hosted centrally at Northwestern and deployed by local CBO staff. Training and coaching of CBO staff on how to use the technology and integrate it into routine HIV testing is provided through capacity building assistance.

Strategy 2 is a "direct-to-consumer" (DTC) model where centralized staff at Northwestern primarily recruit participants nationally through online advertising campaigns and manage participants' engagement. HIV/STI testing kits are shipped directly to YMSM, and upon documentation of an HIV negative test result, participants are delivered KIU! This DTC model has been widely adopted in technology dissemination but it is innovative in terms of implementation of HIV prevention programs.

The investigators will accomplish the goal to inform eHealth intervention implementation with two specific aims:

Aim 1: Compare two implementation strategies using a quasi-experimental trial.

The investigators selected a type III hybrid implementation-effectiveness design, which prioritizes empirical comparison of implementation strategies while also collecting evidence of effectiveness. KIU will be delivered using Strategy 1 (CBOs) in 22 counties for two years; simultaneously, the investigators will deliver KIU nationally using Strategy 2 (DTC). YMSM participants in the DTC strategy will be matched to CBO strategy participants based on post-hoc propensity scores. Implementation and effectiveness outcome data will be collected from YMSM participants, CBOs, and the technology vendor. The primary outcomes are public health impact (defined as reach X effectiveness) and cost per infection averted, a key component of CDC decision making about which HIV prevention programs will be supported. There continues to be equipoise for the trial (i.e., either strategy could be superior). Because implementation success can be defined differently for different stakeholders, the investigators will also continue to collect and report as secondary outcomes multiple metrics of reach, effectiveness, and implementation.

Aim 2: Examine adoption characteristics that explain variability in implementation outcomes.

There is remarkable variability in implementation success when CBOs adopt evidence-based interventions. The investigators will seek to explain variability in implementation success across counties by conducting mixed-methods research on the domains from the consolidated framework for implementation research (CFIR), such as county characteristics, adaptations, support from organization leadership, and approach to planning adoption. Data on CFIR characteristics will be collected through administrative data, surveys, and telephone interviews with key stakeholders.

In addition to these 2 specific aims, the investigators will explore sustainment of KIU! at the completion of the study. CBOs will be provided with materials to facilitate applying for external funding to continue to provide KIU! after study completion, including an Impact Tool to estimate local impact and costs. The investigators will also examine factors that predict applying for funding and ongoing sustainment. For Strategy 2, through consultation with the CDC, capacity building assistance providers, health departments, and small businesses involved in Health 2.0 initiatives, the investigators will examine models for ongoing sustainment of the DTC model.

ELIGIBILITY:
Inclusion Criteria:

* recently received an HIV negative test result OR self-report negative or unknown HIV status
* speaks/reads English
* has an active email address

Exclusion Criteria:

* has not been on PrEP and adherent for 6 months prior

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender men or non-binary
Enrollment: 2125 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Public Health Impact (reach X effectiveness) | 12 Weeks
  Public Health Impact (PHI) involves the reach into the county's YMSM community, weighted by HIV risk (i.e., engagement of YMSM from higher risk communities is valued more), and effectiveness at reducing HIV risk, defined as condomless anal sex, STIs, and adherent PrEP use (i.e., three major risk factors for HIV expected to be modified by KIU!).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Mustanski, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI agrees to develop a de-identified database, codebook, and mechanism by which IPD could be shared with other investigators upon approval of the PI. Data will be available for request approximately 6 months after completion of the project. Interested investigators will be asked to complete a standardized request form stating the specific aims of the analysis, the analytic plans, resources the requestors have to carry out the project, the proposed timeline, and distribution goals (manuscripts and/or grant application). The PI will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to undertake the request, how data will be protected/managed, and whether there are sufficient resources to honor the request. If any of these issues are problematic, the PI will attempt to negotiate a fair resolution with the interested parties and/or with NIH program staff.

REFERENCES:
- [Derived] Zamantakis A, Zapata JP, Smith JD, Danielson EC, Macapagal K, Saber R, Li D, Benbow N, Mustanski B. Incentivizing Prevention: Community Based Organizations' Perceptions on Financial Incentives for Recruitment and Retention of Participants in Keep it Up! (KIU!), an eHealth HIV Prevention Intervention. AIDS Behav. 2025 Nov 21. doi: 10.1007/s10461-025-04963-w. Online ahead of print. PMID 41266922
- [Derived] Mustanski B, Benbow N, Macapagal K, Li D, Madkins K, Saber R, Linas B, Smith JD, Brown CH, Munroe S, Reddy S, Schackman BR, Swann G, Janulis P, Zamantakis A, Zapata JP. Comparing Implementation and Effectiveness Outcomes for Two Implementation Strategies of the Keep It Up! Digital HIV Prevention Program: A Type 3 Hybrid Effectiveness-Implementation Trial. AIDS Behav. 2025 Dec;29(12):4030-4042. doi: 10.1007/s10461-025-04838-0. Epub 2025 Aug 19. PMID 40826259
- [Derived] Zamantakis A, Zapata JP, Greenawalt I, Knapp AA, Benbow N, Mustanski B. Barriers and Facilitators to Implementing Keep It Up!, A Digital Health Intervention, in Community-Based Organizations. AIDS Behav. 2024 Dec;28(12):3944-3955. doi: 10.1007/s10461-024-04525-6. Epub 2024 Oct 10. PMID 39387999
- [Derived] Li DH, Zamantakis A, Zapata JP, Danielson EC, Saber R, Benbow N, Smith JD, Swann G, Macapagal K, Mustanski B. A mixed-methods approach to assessing implementers' readiness to adopt digital health interventions (RADHI). Implement Sci Commun. 2024 Aug 27;5(1):91. doi: 10.1186/s43058-024-00628-2. PMID 39192345